CLINICAL TRIAL: NCT07165639
Title: Association Between Inflammation Biomarkers and Neurocognitive Performance Among Adolescents Living With HIV in Eswatini
Brief Title: The Eswatini Study on Neurocognitive Performance in Adolescents Living With HIV
Status: Not yet recruiting | Type: Observational
Sponsor: Eswatini Nazarene Health Institutions (Other)
Collaborators: Baylor Foundation Eswatini (Unknown)
Responsible Party: Sponsor
Other Study IDs: EHHRRB 049/2025
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: adolescent; Human Immunodeficiency Virus; inflammation biomarkers; neurocognitive performance; Eswatini
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases, HIV positive adolescent: This group comprises adolescents aged 13-19 years living with HIV in Eswatini, recruited from Baylor College of Medicine Children's Foundation-Eswatini Centers of Excellence and affiliated clinical sites. Participants are virally suppressed or on antiretroviral therapy (ART) and will undergo standardized neurocognitive assessments, psychosocial evaluations, and clinical data collection, including CD4+ T-cell count, plasma viral load, ART regimen history, and inflammatory biomarker profiling. No therapeutic or behavioral intervention will be administered as part of the study; all procedures are observational and non-invasive. The objective is to characterize neurocognitive performance and identify biological correlates of cognitive outcomes in adolescents with perinatally acquired HIV.
- Group: HIV-Negative Adolescents: This group consists of adolescents aged 13-19 years who are HIV-negative, recruited from Raleigh Fitkin Memorial (RFM) Hospital in Eswatini. Participants will undergo the same standardized neurocognitive assessments and psychosocial evaluations as their HIV-positive counterparts. No therapeutic or behavioral intervention will be administered; all procedures are observational and non-invasive. This group serves as a control population to facilitate comparative analyses of neurocognitive performance and inflammatory biomarker profiles, thereby helping to isolate the effects of HIV infection on neurodevelopmental outcomes

SUMMARY:
This study explores the link between inflammatory biomarkers and neurocognitive performance in adolescents living with HIV (ALHIV) in Eswatini. Persistent HIV infection during adolescence has been associated with ongoing systemic inflammation and subsequent neurocognitive dysfunction. However, the exact nature of this relationship is not well-defined, especially in resource-limited settings where epidemiological and mechanistic data are scarce.

objectives

* To determine the prevalence of cognitive impairment among a sample of adolescents living with HIV, compared to HIV-negative adolescents in Eswatini
* To assess the relationship between neurocognitive performance and current viral load status in adolescent living with HIV (ALHIV).
* To examine the association between inflammation biomarkers and viral load suppression status in ALHIV.
* To investigate whether adolescents with HIV experiencing neurocognitive decline exhibit a high inflammatory status.

A case-control design will be employed, involving 80 adolescents aged 13-19 years: 50 who are HIV-positive and 30 HIV-negative controls. Participants will be recruited from Baylor Manzini and Mbabane, as well as Raleigh Fitkin Memorial Hospital. Neurocognitive function will be evaluated using the Symbol Digit Modalities Test, focusing on areas such as processing speed, motor coordination, attention, and visual scanning.

Blood samples will be collected to measure key inflammatory biomarkers, including C-reactive protein (CRP), soluble CD14 (sCD14), lipopolysaccharide (LPS), soluble CD163 (sCD163), and monocyte chemoattractant protein-1 (MCP-1). Sociodemographic and clinical data will be gathered through questionnaires and medical record reviews.

Primary outcomes will include neurocognitive performance scores, while secondary outcomes will involve biomarker levels and their correlation with cognitive function. Multivariate regression models will assess associations, adjusting for confounders such as age, sex, education, and HIV disease severity. Structural equation modeling will be used to explore potential mediators in the inflammation-cognition pathway.

DETAILED DESCRIPTION:
Adolescents living with HIV (ALHIV) in sub-Saharan Africa face a complex health burden that goes beyond virological control. In Eswatini, where HIV prevalence ranks among the highest globally, the combination of chronic infection, immune dysregulation, and neurodevelopmental vulnerability poses a significant public health challenge. Although antiretroviral therapy (ART) has greatly improved survival rates, emerging evidence indicates that ongoing immune activation may lead to subtle yet clinically significant neurocognitive deficits in youth. These impairments can impact academic performance, psychosocial functioning, and long-term quality of life.

This study aims to explore the biological correlates of neurocognitive performance in ALHIV, with a particular focus on inflammatory biomarkers. It seeks to determine the extent to which systemic inflammation measured through specific immunological markers relates to cognitive functioning in adolescents and whether these associations differ between HIV-positive and HIV-negative individuals.

Utilizing a case-control design, the study will generate comparative data to enhance understanding of the neuroimmune interface in this population. Study Population and Recruitment The study will enroll 80 adolescents aged 13 to 19 years, consisting of: 50 HIV-positive participants, recruited from HIV care centers at Baylor College of Medicine Children's Foundation-Eswatini (Manzini & Mbabane), and Raleigh Fitkin Memorial Hospital. 30 HIV-negative controls, matched by age and sex, recruited from the same geographic catchment areas to ensure contextual comparability. Eligibility criteria include confirmed HIV status (positive or negative), age within the specified range, and capacity to participate in neurocognitive testing. Exclusion criteria include acute illness, neurological disorders unrelated to HIV, or inability to provide informed consent/assent.

Neurocognitive Assessment Protocol Cognitive functioning will be assessed using the Symbol Digit Modalities Test (SDMT), a standardized neuropsychological instrument sensitive to changes in processing speed and attention. The SDMT is particularly suitable for use in low-resource settings due to its minimal language dependence and brief administration time. It evaluates: Visual scanning Psychomotor speed Sustained attention Working memory Testing will be conducted in a quiet, controlled environment by trained research personnel fluent in local languages and familiar with adolescent developmental norms.

Biomarker Collection and Analysis Venous blood samples will be collected from all participants under sterile conditions. Samples will be processed and stored according to biosafety protocols and analyzed using enzyme-linked immunosorbent assay (ELISA) techniques. The following biomarkers will be quantified: C-reactive protein (CRP): A general marker of systemic inflammation. Soluble CD14 (sCD14): Reflects monocyte activation and microbial translocation. Lipopolysaccharide (LPS): Indicates gut barrier dysfunction and endotoxemia. Soluble CD163 (sCD163): Associated with macrophage activation and neurodegeneration. Monocyte chemoattractant protein-1 (MCP-1): A chemokine involved in leukocyte recruitment and neuroinflammatory signaling. These biomarkers were selected based on their relevance to HIV-associated immune activation and their potential role in neurocognitive outcomes.

Sociodemographic and Clinical Data Collection

Participants will engage in structured interviews and complete questionnaires to gather sociodemographic information, including:

* Age
* Gender
* Educational attainment
* Household composition
* Socioeconomic status

Clinical data will be sourced from medical records, encompassing:

* Duration of HIV infection
* ART regimen and adherence history
* CD4+ T-cell count and viral load
* History of opportunistic infections
* Neurological symptoms or diagnoses This comprehensive dataset will facilitate robust adjustment for confounding variables in statistical analyses.

Outcome Measures

Primary Outcome:

Neurocognitive performance scores derived from SDMT results.

Secondary Outcomes:

* Quantitative levels of inflammatory biomarkers.
* Correlation coefficients between biomarker levels and cognitive scores.
* Group differences in biomarker profiles and cognitive outcomes. Statistical Analysis Plan

Data will be analyzed using multivariate regression models to evaluate the relationship between inflammatory biomarkers and neurocognitive performance. These models will adjust for potential confounders, including:

* Age
* Sex
* Educational level
* HIV disease severity (e.g., CD4 count, viral load)
* ART adherence Interaction terms will be explored to determine if the strength of associations varies by HIV status. Additionally, structural equation modeling (SEM) will be employed to investigate potential mediating pathways, such as the role of monocyte activation in linking HIV infection to cognitive impairment. SEM allows for the simultaneous estimation of direct and indirect effects, providing a nuanced understanding of the biological mechanisms involved.

Ethical Considerations The study protocol has been reviewed and approved by the Eswatini Health and Human Research Review Board (EHHRRB). Informed consent will be obtained from all participants aged 18 and above, and assent will be obtained from minors alongside parental or guardian consent. All data will be anonymized and securely stored, with access restricted to authorized personnel. Participants will be informed of their right to withdraw at any time without consequence.

Data Management and Quality Assurance Data will be entered into a secure electronic database with built-in validation checks. Double data entry and periodic audits will be conducted to ensure accuracy. Laboratory assays will be performed in duplicate, and inter-assay variability will be monitored. All research staff will undergo training in Good Clinical Practice (GCP) and ethical conduct of research involving human subjects.

Potential Risks and Benefits Risks to participants are minimal and primarily related to blood draw procedures (e.g., discomfort, bruising). Psychological distress from cognitive testing is considered low. Participants may benefit from increased awareness of their cognitive health and receive referrals for further evaluation if significant impairments are detected.

Significance and Innovation

This study addresses a critical gap in understanding HIV-associated neurocognitive impairment in adolescents, particularly in high-prevalence, resource-limited settings. By integrating immunological and neuropsychological data, it offers a novel approach to characterizing the neuroimmune interface in ALHIV. The findings may:

* Identify biomarkers predictive of cognitive decline.
* Inform early screening and intervention strategies.
* Support the development of targeted therapies to mitigate neuroinflammation.
* Enhance clinical guidelines for adolescent HIV care. Moreover, the study contributes to global efforts to improve the long-term outcomes of adolescents living with HIV, aligning with UNAIDS goals for health equity and sustainable development.

ELIGIBILITY:
Inclusion Criteria:

* Cases

  * Adolescents aged 13-19 years
  * HIV-positive
  * Undergoing antiretroviral therapy at Baylor Clinic
  * Providing consent or assent to participate

Controls

* Adolescents aged 13-19 years
* HIV-negative
* Providing consent or assent to participate

Exclusion Criteria:

* Exclusion Criteria

  * Recent (within 2 months) acute conditions: influenza, COVID-19, TB, acute gastroenteritis (as these conditions elevate CRP levels)
  * Chronic conditions: diabetes, hypertension, asthma
  * Neurological disorders: epilepsy, cerebrovascular accident, neurodegenerative diseases
  * History of significant cranial trauma or perinatal complications
  * All the aforementioned conditions will be identified through self-reported data and medical records.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population will encompass all adolescents attending RFM hospitals, Baylor RFM, and Baylor Mbabane: 1. Adolescents aged 13 to 19 years who are on antiretroviral therapy (ART) and attending the Baylor clinic at RFM and Baylor Mbabane. 2. HIV-negative adolescents aged 13 to 19 years who meet the inclusion criteria and are consulting at the RFM hospital outpatient department.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Neurocognitive performance | baseline
  The Symbol Digit Modalities Test (SDMT) assesses neurocognitive performance by evaluating processing speed, attention, and visual-motor coordination. Participants are required to use a key to match symbols with digits as swiftly as possible within a 90-second timeframe, with the score indicating the number of correct matches. Z-scores, which typically range from -3.0 to +3.0, are employed to interpret results in relation to age and population norms. A score of 0 denotes average performance, while scores between +1 and +3 suggest above-average cognitive abilities. Conversely, scores from -1 to -1.5 may indicate mild impairment, and those below -1.5 often highlight clinically significant deficits, particularly in adolescents.

SECONDARY OUTCOMES:
Quantitative levels of inflammatory biomarkers. | baseline
  Blood samples will be collected to assess inflammatory biomarkers, including CRP, sCD14, LPS, sCD163, and MCP-1. The typical interpretation of their levels is as follows:
  CRP (C-reactive protein)
  * Low: <1 mg/L
  * Normal: 1-3 mg/L
  * High: >3 mg/L sCD14 (soluble CD14)
  * Low: <1000 ng/mL
  * Normal: 1000-1500 ng/mL
  * High: >1500 ng/mL LPS (lipopolysaccharide)
  * Low: <0.05 EU/mL
  * Normal: 0.05-0.1 EU/mL
  * High: >0.1 EU/mL sCD163 (soluble CD163)
  * Low: <1000 ng/mL
  * Normal: 1000-2000 ng/mL
  * High: >2000 ng/mL MCP-1 (monocyte chemoattractant protein-1)
  * Low: <100 pg/mL
  * Normal: 100-200 pg/mL
  * High: >200 pg/mL These ranges may vary slightly depending on the assay used and the population studied, but they provide a general framework for interpreting inflammatory status.

CONTACTS AND LOCATIONS:
Overall Officials: Phathizwe M Mantshana, BSc, Principal Investigator — Eswatini Nazarene Health Institution; Sarah H Perry, Ass professor, Study Director — Baylor College of Medicine; Debrah Vambe, MD, Study Director — Baylor College of Medicine; Mkunde S Chachage, PHD, Study Director — University of Dar es Salaam-Mbeya; Clement Gascua AduGyamfi, G AduGyamfi,, PHD, Study Director — Baylor College of Medicine; Alfred Balasa,, Associate Professor, Study Director — Texas Children's Hospital Austin Baylor College of Medicine; ANDREW R DINARDO, associate professor, Study Director — Baylor College of Medicine
Locations (1):
- Eswatini Nazarene Health Institution, Baylor College of Medicine Children's Foundation-Eswatini (Centers of Excellence in Mbabane and satellite clinic in Manzini in Raleigh Fitkin Memorial Hospital), Manzini, Eswatini

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) to be shared will include fully de-identified datasets derived from standardized neurocognitive assessments, core demographic variables (such as age, biological sex, and educational attainment), HIV-specific clinical indicators (e.g., CD4+ T-cell count, plasma viral load, and antiretroviral therapy regimen), and validated psychosocial measures collected throughout the study. All direct and indirect identifiers will be removed in accordance with international data protection standards and ethical research practices, ensuring participant confidentiality. The availability of these IPD will facilitate rigorous secondary analyses focused on neurocognitive functioning among adolescents living with HIV, thereby contributing to the broader scientific understanding of HIV-associated neurodevelopmental trajectories. The study protocol and statistical analysis plan will be made publicly accessible via ClinicalTrials.gov.
Supporting Information: Study Protocol, SAP
Time Frame: Data from this study will be made available beginning six months after the primary publication of results.
Access Criteria: Anonymized individual participant data will be made available to qualified members of the scientific community in accordance with the Baylor Foundation Eswatini data sharing policy. Access will be granted upon formal request and subject to review and approval procedures designed to ensure ethical use, data security, and alignment with participant consent provisions.

REFERENCES:
- [Background] Swanta N, Aryal S, Nejtek V, Shenoy S, Ghorpade A, Borgmann K. Blood-based inflammation biomarkers of neurocognitive impairment in people living with HIV. J Neurovirol. 2020 Jun;26(3):358-370. doi: 10.1007/s13365-020-00834-3. Epub 2020 Mar 19. PMID 32193795
- [Background] Moschopoulos CD, Stanitsa E, Protopapas K, Kavatha D, Papageorgiou SG, Antoniadou A, Papadopoulos A. Multimodal Approach to Neurocognitive Function in People Living with HIV in the cART Era: A Comprehensive Review. Life (Basel). 2024 Apr 15;14(4):508. doi: 10.3390/life14040508. PMID 38672778
- [Background] Mouchati C, El Kamari V, Sattar A, Yu J, McComsey GA. Comprehensive assessment of neurocognitive function, inflammation markers, and adiposity in treated HIV and control. Medicine (Baltimore). 2022 Oct 21;101(42):e31125. doi: 10.1097/MD.0000000000031125. PMID 36281153
- [Background] Kapetanovic S, Giganti MJ, Abzug MJ, Lindsey JC, Sirois PA, Montepiedra G, Canniff J, Agwu A, Boivin MJ, Weinberg A; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) network. Plasma biomarker factors associated with neurodevelopmental outcomes in children with perinatal HIV infection and controlled viremia. AIDS. 2021 Jul 15;35(9):1375-1384. doi: 10.1097/QAD.0000000000002862. PMID 33710019
- [Background] Hoare J, Myer L, Heany S, Fouche JP, Phillips N, Zar HJ, Stein DJ. Cognition, Structural Brain Changes, and Systemic Inflammation in Adolescents Living With HIV on Antiretroviral Therapy. J Acquir Immune Defic Syndr. 2020 May 1;84(1):114-121. doi: 10.1097/QAI.0000000000002314. PMID 32032303
- [Background] Anderson AM, Jang JH, Easley KA, Fuchs D, Gisslen M, Zetterberg H, Blennow K, Ellis RJ, Franklin D, Heaton RK, Grant I, Letendre SL. Cognitive and Neuronal Link With Inflammation: A Longitudinal Study in People With and Without HIV Infection. J Acquir Immune Defic Syndr. 2020 Dec 15;85(5):617-625. doi: 10.1097/QAI.0000000000002484. PMID 32932412
- See also: Peer-reviewed article in Journal of NeuroVirology (2020) identifying blood-based inflammatory biomarkers-such as CCL8, TIMP-1, and IL-23-associated with neurocognitive impairment in people living with HIV, using multivariate regression analysis — https://doi.org/10.1007/s13365-020-00834-3
- See also: Peer-reviewed article in Medicine (Baltimore) (2022) examining associations between inflammatory biomarkers and neurocognitive function in people living with HIV, highlighting links between systemic inflammation and cognitive impairment. — https://doi.org/10.1097/md.0000000000031125
- See also: This study investigates how plasma biomarkers-such as sCD14, IL-6, and TNF-α-correlate with neurodevelopmental outcomes in children with perinatal HIV who are virally suppressed. It's a key reference for understanding the biological mechanisms underlying — https://journals.lww.com/aidsonline/abstract/2021/07150/plasma_biomarker_factors_associated_with.5.aspx
- See also: Peer-reviewed article from the *Journal of NeuroVirology* (2020) examining how earlier antiretroviral therapy initiation in youth with vertically transmitted HIV is associated with improved brain structure and working memory-related neural activation. — https://infospace.mrc.ac.za/bitstreams/4588c400-a2e8-4f56-9ca4-d9e4dc1dd68a/download
- See also: ClinicalTrials.gov protocol entry for "The Eswatini Study on Neurocognitive Performance in Adolescents Living With HIV," detailing study identification, design, outcome measures, data sharing plans, and references for related publications and supporting — https://discovery.ucl.ac.uk/id/eprint/10110682/